CLINICAL TRIAL: NCT06902129
Title: Engineering Evaluation of Aerosol Flow, Inhalation Pattern Control, and Digital Accuracy in Three Breath-Activated EDDIS Systems (VMT, Atomizer, Ultrasonic) Using Inert NaCl-Based Formulation With Chitosan Nanoparticles
Brief Title: Validation of Safety and Performance of Three EDDIS Breath-Activated Portable Inhalation Systems
Acronym: EDDIS-ENG
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Petrov, Andrey (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Device Feasibility
Other Study IDs: EDDIS-ENG-03D
Record Dates: First submitted 2025-03-21; First posted 2025-03-30 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Healthy Volunteers; Drug Delivery Systems; Inhalation of Liquid Air; Administration Site Injury
Keywords: Breath-Activated Inhaler; Aerosol Delivery; Drug Delivery Device; Portable Inhaler; Inhalation Therapy; Bioavailability
MeSH Terms: interventions — Nebulizers and Vaporizers; Ultrasonography

STUDY DESIGN:
Intervention Model Description: Crossover Assignment
Masking Description: None (Open Label)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Healthy Volunteers - VMT First (Experimental): All participants receive the VMT device first, followed by the Atomizer and Ultrasonic devices in a randomized crossover sequence using a non-active saline aerosol with chitosan nanoparticles. Device performance parameters and user tolerability will be recorded
  Interventions: Device: EDDIS Platform - Portable Inhalation Delivery Systems (VMT, Atomizer, Ultrasonic)
- Healthy Volunteers - Atomizer First (Experimental): All participants receive the Atomizer device first, followed by the VMT and Ultrasonic devices in a randomized crossover sequence using a non-active saline aerosol with chitosan nanoparticles. Device performance parameters and user tolerability will be recorded
  Interventions: Device: EDDIS Platform - Portable Inhalation Delivery Systems (VMT, Atomizer, Ultrasonic)
- Healthy Volunteers - Ultrasonic First (Experimental): All participants receive the Ultrasonic device first, followed by the VMT and Atomizer devices in a randomized crossover sequence using a non-active saline aerosol with chitosan nanoparticles. Device performance parameters and user tolerability will be recorded
  Interventions: Device: EDDIS Platform - Portable Inhalation Delivery Systems (VMT, Atomizer, Ultrasonic)

INTERVENTIONS:
Device: EDDIS Platform - Portable Inhalation Delivery Systems (VMT, Atomizer, Ultrasonic) — A set of three single-use, disposable, closely matched and uniform in size, breath-actuated, digitally monitored portable inhalation devices designed for precision aerosol delivery. Devices include a vibrating mesh (VMT), an atomizer-based unit (ATM), and an ultrasonic micro-vibration unit (ULT). Each system records inhalation parameters and connects via Bluetooth to a mobile application for real-time feedback and logging. Used to assess technical performance, gas dynamics, and digital control functions using a non-active NaCl-based aerosol with chitosan nanoparticles.
  Other Names: EDDIS-VMT, EDDIS-ATM, EDDIS-ULT, Breath-actuated Inhaler, Disposable Digital Inhalation Device

SUMMARY:
This is a crossover study to evaluate real-time performance, airflow control, user-device interaction, and safety systems of three portable inhalation systems from the EDDIS platform. The formulation is non-pharmacological and inert.

Each volunteer will use all three devices in random order. Primary endpoints focus on gas dynamics, inhalation recording accuracy, device integrity, and user tolerability.

DETAILED DESCRIPTION:
This is a device-only evaluation of three portable inhalation delivery systems from the EDDIS platform (VMT, Atomizer, Ultrasonic). The study focuses on technical performance, gas dynamics, safety system integrity, and user-device interaction under controlled conditions in healthy adult volunteers.

Each device is breath-actuated, disposable, and digitally integrated with a smartphone application. The inhaled formulation consists of sterile 0.9% sodium chloride containing suspended chitosan nanoparticles (<200 nm), designed to simulate complex aerosol behavior without delivering any active pharmaceutical ingredients.

The study employs a crossover design, allowing each subject to evaluate all three devices in a randomized sequence. Performance characteristics such as airflow resistance, aerosol output, inspiratory detection sensitivity, power consumption, and digital logging accuracy will be assessed. Special emphasis is placed on safety-related engineering features, including detection of abnormal inhalation patterns (e.g., cough-like events), child-lock functionality, and plume behavior under variable user conditions.

This study does not involve any drug or therapeutic intervention, is not classified as a clinical investigation under EU MDR or Swissmedic regulations, and does not require ethics committee oversight. The primary objective is to validate the EDDIS platform as a modular, scalable, and precisely controlled aerosol delivery system suitable for further development in both clinical and non-clinical applications.

ELIGIBILITY:
Inclusion Criteria:

Age between 21 and 75 years

* Generally healthy adult (no known systemic or chr
* Normal pulmonary function (FEV1 ≥ 80% predicted at screening)
* Body Mass Index (BMI) between 18.5 and 30 kg/m²
* Able and willing to provide written informed consent form
* Current or prior use of tabac

Exclusion Criteria:

* Body temperature ≥ 38.0°C on the day of screening or inhalation
* Acute respiratory infection, cough, cold, or any inflammatory disease of the head and neck within the last 2 weeks
* History of asthma, COPD, or other chronic pulmonary disease
* History of thoracic or lung surgery
* Known cardiovascular pathology, including uncontrolled or progressive hypertension
* Pulmonary bleeding, hemoptysis, or blood in saliva
* Diagnosed emphysema
* Known bleeding disorders or use of anticoagulants
* Known allergy or hypersensitivity to chitosan or related compounds
* Any inhalation-induced adverse reactions during baseline assessment (e.g., cough reflex not resolving within 30 seconds)
* Use of investigational drugs or participation in another clinical study within 30 days prior to enrollment
* Unwillingness or inability to follow the study plan or to comply with the requirements of the informed consent agreement
* Any condition which, in the opinion of the investigator, may interfere with study participation or result interpretation

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-11-09 (Estimated); Primary Completion 2026-03-10 (Estimated); Study Completion 2026-04-12 (Estimated)

PRIMARY OUTCOMES:
Airflow Resistance Measurement | up to 72 hours
  change in airflow resistance (cmH₂O/L/s) across three devices (cmH₂O/L/s via digital sensor output)
Inspiratory Flow Detection Accuracy | up to 72 hours
  quantitative indicators (%) of detection of valid inhalation efforts compared to reference pneumotachograph

SECONDARY OUTCOMES:
Device Recording Fidelity | up to 6 hours (during all sessions)
  rate of accurate digital logging of breath events ( accuracy vs manually annotated data) %)
Subjective Device Comfort Score | up to 6 hours (after each device use - 3 total sessions)
  self-reported comfort level assessed immediately after using each device, using a standardized 10-point Visual Analog Scale (VAS), where 0 represents "very uncomfortable" and 10 represents "extremely comfortable"
Safety Event Detection | up to 3 hours (during each inhalation session per device)
  The number of abnormal inspiratory events detected per device, including simulated coughs, breath holding, or irregular inspiratory flow patterns. Events are automatically logged by the digital security system and manually reviewed

CONTACTS AND LOCATIONS:
Locations (1):
- Central Contact, Lausanne, Switzerland